CLINICAL TRIAL: NCT02263079
Title: A Phase IIIb, Randomized, Open-Label Study of Pegylated Interferon Alfa-2A in Combination With Lamivudine or Entecavir Compared With Untreated Control Patients in Children With HBeAg Positive Chronic Hepatitis B in the Immune-Tolerant Phase
Brief Title: A Study of Pegylated Interferon Alfa-2A in Combination With Lamivudine or Entecavir Compared With Untreated Control Group in Children With Hepatitis B Envelope Antigen (HBeAg)-Positive Chronic Hepatitis B (CHB) in the Immune-Tolerant Phase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV25361; 2006-000977-31 (EudraCT Number)
Record Dates: First submitted 2014-10-02; First posted 2014-10-13 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Pediatric Immuno-Tolerant Chronic Hepatitis B
MeSH Terms: interventions — entecavir; Lamivudine; peginterferon alfa-2a

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Peg-IFN-Alfa-2A + Lamivudine or Entecavir (Experimental): Participants will receive lamivudine or entecavir alone for 8 weeks followed by peg-IFN-alfa-2A in combination with lamivudine or entecavir for 48 weeks.
  Interventions: Drug: Entecavir; Drug: Lamivudine; Drug: Pegylated Interferon Alfa-2A
- Untreated Control Participants (No Intervention): Untreated control participants will be observed up to 80 weeks.
- Peg-INF-Alfa-2A Monotherapy (Experimental): Participants will receive Peginterferon Alfa 2A subcutaneously once weekly with dosing based on body surface area (BSA) categories for 48 weeks.
  Interventions: Drug: Pegylated Interferon Alfa-2A

INTERVENTIONS:
Drug: Entecavir — Participants will receive entecavir, either as a film-coated tablet or oral solution, once daily at a dose of 0.015 milligrams per kilogram (mg/kg) (maximum daily dose of 0.5 mg).
  Arms: Peg-IFN-Alfa-2A + Lamivudine or Entecavir
Drug: Lamivudine — Participants will receive lamivudine, either as a film-coated tablet or oral solution, once daily at a dose of 3 mg/kg (maximum daily dose of 100 mg).
  Arms: Peg-IFN-Alfa-2A + Lamivudine or Entecavir
Drug: Pegylated Interferon Alfa-2A — Participants will receive pegylated interferon-alfa-2A at a body surface area (BSA) based dose of 180 micrograms per 1.73 square meter (mcg/1.73m^2) BSA.
  Other Names: Pegasys, Peg-IFN-Alfa-2A
  Arms: Peg-IFN-Alfa-2A + Lamivudine or Entecavir; Peg-INF-Alfa-2A Monotherapy

SUMMARY:
This randomized, controlled, parallel group, open-label multicenter study will evaluate the efficacy and safety of a combination of pegylated interferon alfa-2A (Pegasys) plus lamivudine or entecavir compared with an untreated control group in participants with HBeAg positive CHB in the immune tolerant phase. NOTE: STUDY RECRUITMENT HAS BEEN TERMINATED

ELIGIBILITY:
Inclusion Criteria:

* Positive for HBsAg and HBeAg for more than 6 months prior to baseline
* Detectable HBV-DNA (>20,000 IU/mL) as measured by polymerization chain reaction (PCR) or hybridization on at least 2 occasions at least one month apart with the latest determination obtained less than or equal to (</=) 42 days prior to baseline
* Compensated liver disease (Child-Pugh Class A clinical classification)
* Either Liver biopsy performed within 2 years prior to baseline showing no or minimal fibrosis (Liver Biopsy Scores and stable normal ALT levels (less than or equal to upper limit of normal [ULN]) during the 6 months leading up to baseline (including two separate occasions at least 1 month apart over the 6 months prior to baseline). Screening ALT levels must be normal (</= ULN) OR Stable normal ALT levels (</= ULN), during the 1 year leading up to baseline (including three separate occasions at least 1 month apart over the 1 year prior to baseline) and no signs of hepatocellular carcinoma (HCC), advanced fibrosis/cirrhosis, or splenomegaly on liver abdominal ultrasound at screening. Screening ALT levels must be normal (</= ULN)

Exclusion Criteria:

* Participants who have received investigational drugs or licensed treatments with anti HBV activity (Exception: Participants who have had a limited [</= 7-day] course of acyclovir for herpetic lesions more than 1 month before the study baseline visit are not excluded)
* Participants who have participated in any other clinical trial or who have received any investigational drug within 6 months prior to baseline
* Known hypersensitivity to interferon (IFN), pegylated interferon-alfa-2a or lamivudine or entecavir
* Positive test results at screening for hepatitis A virus Immunoglobulin M (IgM) antibody (Ab), anti-hepatitis C virus (HCV) Ab, anti- hepatitis D (HDV) Ab or anti-human immunodeficiency virus (HIV) Ab
* Decompensated liver disease (e.g., Child-Pugh Class B or C clinical classification or clinical evidence such as ascites or varices)
* Advanced fibrosis or cirrhosis
* Suspicion of HCC on liver abdominal ultrasound (all patients to have liver abdominal ultrasound within 6 months prior to baseline)
* History or other evidence of a medical condition associated with chronic liver disease other than CHB including metabolic liver diseases such as hemochromatosis, Wilson's disease or alpha-1 anti-trypsin deficiency
* Active substance abuse within 6 months prior to screening
* Sexually active females of childbearing potential and sexually active males who are not willing to utilize reliable contraception during treatment and for 90 days following the end of treatment
* Females who are pregnant or who are breastfeeding (females of childbearing potential who have a positive urine or serum pregnancy test result within 24 hours of baseline are excluded)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- United States (3):
  - Children's Mercy Hosp Clinics, Kansas City, Missouri
  - Columbia University, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Womens and Childrens Hospital; Department of Gastroenterology, North Adelaide, South Australia, Australia
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Gent, Ghent
- Germany (4):
  - Universitätsklinikum Essen; Klinik für Kinder- und Jugendmedizin Pädiatrie II, Essen
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Zentrum für Kinder- und Jugendmedizin, Mainz
  - Dr. von Haunerschen Kinderspital, Kinderchirurgische Klinik und Poliklinik, München
  - HELIOS Klinikum Wuppertal, Zentrum für Kinder- und Jugendmedizin, Universität Witten-Herdecke, Wuppertal
- Azienda Ospedaliero-Universitaria Policlinico S. Orsola Malpighi; U.O. Malattie Infettive, Bologna, Emilia-Romagna, Italy
- University Malaya Medical Center; Department of Paediatrics, Kuala Lumpur, Malaysia
- Grigore Alexandrescu Emergency Clinical Hospital for Children, Bucharest, Romania
- Russia (2):
  - FSI Scientific research Institute of children's infections, Saint Petersburg
  - MC Gepatolog, Samara
- Chang-Gung Memorial Hospital-Linkou; Division of Pediatric Gastroenterology, Dept Pediatrics, Taoyuan, Taiwan
- Turkey (Türkiye) (4):
  - Cukurova University Medical School Department of Pediatrics; Pediatric Infectious Diseases, Adana
  - Ankara University School of Medicine, Pediatrics Department; Pediatric Gastroenterology, Ankara
  - Hacettepe Uni , School of Medicine; Gastroenterology, Ankara
  - Gazi Universitesi Tip Fakultesi Pediyatri Anabilim Dalı; Pediyatrik Gastroenteroloji, Ankara
- SI Institute of the pediatrics, obstetrics and gynecology, Kyiv, Ukraine
- United Kingdom (4):
  - Birmingham Children'S Hopsital; Liver Unit, Birmingham
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Kings College Hospital NHS Foundation Trust, London
  - North Manchester General Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began as a single-site, three arm IST and was subsequently adapted as a multi-center, two arm study, conducted at 22 sites in Malaysia, Taiwan, Australia, Belgium, Germany, United Kingdom, Italy, Romania, Russian Federation, Turkey, Ukraine and the U.S. Enrolment was stopped prematurely, at which time 62 participants had been enrolled.
Groups:
- Peg-IFN-Alfa-2A + Lamivudine or Entecavir: Participants received lamivudine or entecavir alone for 8 weeks followed by peg-IFN-alfa-2A in combination with lamivudine or entecavir for 48 weeks.
- Untreated Control Participants: Untreated control participants were observed up to 80 weeks.
- Peg-INF-Alfa-2A Monotherapy: Participants received Peginterferon Alfa 2A subcutaneously once weekly with dosing based on body surface area (BSA) categories for 48 weeks.
Period: Overall Study
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants | Peg-INF-Alfa-2A Monotherapy
Started | 26 | 33 | 3
Completed | 23 | 25 | 3 (Completed study but not included in the analysis)
Not Completed | 3 | 8 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 0

BASELINE CHARACTERISTICS:
Population: Due to the low participant number (n=3) in the Peg-INF-Alfa-2A Monotherapy arm, data is not presented in this summary for this arm to avoid participant re-identification as well as in consideration of any summary statistics would be misleading, therefore the three participants were presented in listings in the study report.
Groups:
- Total: Total of all reporting groups
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants | Peg-INF-Alfa-2A Monotherapy | Total
Number analyzed (Participants) | 26 | 33 | 3 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Due to the low participant number (n=3) in the Peg-INF-Alfa-2A Monotherapy arm, data is not presented in this summary for this arm in consideration to avoid participant re-identification.
  Years
    number analyzed (Participants) | 26 | 33 | 0 | 59
    (all) | 11.9 (3.2) | 10.9 (3.7) |  | 11.3 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to the low participant number (n=3) in the Peg-INF-Alfa-2A Monotherapy arm, data is not presented in this summary for this arm in consideration to avoid participant re-identification.
  Participants
    number analyzed (Participants) | 26 | 33 | 0 | 59
    Female | 16 | 14 |  | 30
    Male | 10 | 19 |  | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Due to the low participant number (n=3) in the Peg-INF-Alfa-2A Monotherapy arm, data is not presented in this summary for this arm in consideration to avoid participant re-identification.
  Participants
    number analyzed (Participants) | 26 | 33 | 0 | 59
    Hispanic or Latino | 1 | 0 |  | 1
    Not Hispanic or Latino | 25 | 33 |  | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Due to the low participant number (n=3) in the Peg-INF-Alfa-2A Monotherapy arm, data is not presented in this summary for this arm in consideration to avoid participant re-identification.
  Participants
    number analyzed (Participants) | 26 | 33 | 0 | 59
    Asian | 11 | 11 |  | 22
    Black or African American | 4 | 2 |  | 6
    Multiple | 2 | 0 |  | 2
    Other | 0 | 3 |  | 3
    White | 9 | 17 |  | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Loss of Hepatitis B Surface Antigen (HBsAg) at 24 Weeks Post-End of Treatment/End of Untreated Observation
Description: This endpoint is defined as loss of HBsAg at 24 weeks post-treatment (follow-up Week 24)/end of untreated observation (Week 80). The percentage of responders (response rate) and 95% CI (using the Clopper-Pearson method) for the response rate are presented for each group.
Time Frame: 24 weeks post-treatment/at the end of untreated observation (Week 80)
Population: The Intent to treat (ITT) population was defined as all participants who received at least one dose of study medication of treated group. For untreated group, the ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants
Number analyzed (Participants) | 26 | 33
Percentage of Participants | 3.8 [0.10 to 19.64] | 0 [0.00 to 10.58]

2. Secondary Outcome: Percentage of Participants With Loss of HBsAg
Description: This endpoint is defined as loss of HBsAg at 1 year post-treatment in the treated group. The 95% Confidence Interval of response rate is calculated by Clopper-Pearson method.
Time Frame: 1 year post-end of treatment (End of treatment = Week 56)
Population: The analysis population included participants from the Peg-INF-Alfa-2A arm, who received at least one dose of study medication of treated group. None of the participants from the untreated group were assessed at 1 year post-end of treatment as they were only observed up to 80 weeks (=24 weeks post-treatment for treated participants).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir
Number analyzed (Participants) | 26
Percentage of Participants | 3.8 [0.10 to 19.64]

3. Secondary Outcome: Percentage of Participants With Loss of Hepatitis B Virus Envelope Antigen (HBeAg)
Description: This endpoint is defined as loss of HBeAg at 24 weeks post-treatment (follow-up Week 24)/end of untreated observation (Week 80) and at 1 year post-end of treatment in the treated group. The 95% Confidence Interval of response rate is calculated by Clopper-Pearson method.
Time Frame: 24 weeks post-treatment /end of untreated observation (Week 80), and 1 year post-end of treatment (End of treatment = Week 56)
Population: All participants who received at least one dose of study medication of treated group, and all randomized participants in the untreated group. None of the participants from the untreated group were assessed at 1 year post-end of treatment as they were only observed up to 80 weeks (=24 weeks post-treatment for treated group)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants
Number analyzed (Participants) | 26 | 33
Percentage of Participants
  24 Weeks post-treatment/Week 80 | 3.8 [0.10 to 19.64] | 12.1 [3.40 to 28.20]
  1 year post-end of treatment: number analyzed (Participants) | 26 | 0
  1 year post-end of treatment | 11.5 [2.45 to 30.15] |

4. Secondary Outcome: Percentage of Participants With Seroconversion to Hepatitis B Surface Antibody (Anti-HBs), Defined as Loss of HBsAg and Presence of Anti-HBs
Description: This endpoint measures the seroconversion to anti-HBs defined as loss of HBsAg and presence of anti-HBs at 24 weeks post-treatment (follow-up Week 24)/end of untreated observation (Week 80) and at 1 year post-end of treatment in the treated group. The 95% Confidence Interval of response rate is calculated by Clopper-Pearson method.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants
Number analyzed (Participants) | 26 | 33
Percentage of Participants
  24 Weeks post-treatment/Week 80 | 3.8 [0.10 to 19.64] | 0.0 [0.00 to 10.58]
  1 year post-end of treatment: number analyzed (Participants) | 26 | 0
  1 year post-end of treatment | 3.8 [0.10 to 19.64] |

5. Secondary Outcome: Percentage of Participants With Seroconversion to Hepatitis B Envelope Antibody (Anti-HBe), Defined as Loss of HBeAg and Presence of Anti-HBe
Description: This endpoint measures the seroconversion to anti-HBe defined as loss of HBeAg and presence of anti-HBe at 24 weeks post-treatment (follow-up Week 24)/end of untreated observation (Week 80) and at 1 year post-end of treatment in the treated group. The 95% Confidence Interval of response rate is calculated by Clopper-Pearson method.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants
Number analyzed (Participants) | 26 | 33
Percentage of Participants
  24 Weeks post-treatment/Week 80 | 0.0 [0.00 to 13.23] | 9.1 [1.92 to 24.33]
  1 year post-end of treatment: number analyzed (Participants) | 26 | 0
  1 year post-end of treatment | 7.7 [0.95 to 25.13] |

6. Secondary Outcome: Percentage of Participants With Different Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Levels (Less Than [<] 20,000 International Units Per Milliliter [IU/mL], < 2000 IU/mL, or Undetectable HBV DNA)
Description: This endpoint measures different HBV DNA levels (<20000 IU/mL, <2000 IU/mL and undetectable) measured by PCR or hybridization at 24 weeks post-treatment (follow-up Week 24)/end of untreated observation (Week 80) and at 1 year post-treatment in the treated group. HBV-DNA undetectable is defined as <29 IU/mL. The 95% Confidence Interval of response rate is calculated by Clopper-Pearson method.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants
Number analyzed (Participants) | 26 | 33
Percentage of Participants
  HBV-DNA <20000 IU/mL at follow up Week 24/Week 80 | 7.7 [0.95 to 25.13] | 12.1 [3.40 to 28.20]
  HBV-DNA <2000 IU/mL at follow up Week 24/Week 80 | 7.7 [0.95 to 25.13] | 12.1 [3.40 to 28.20]
  HBV-DNA Undetectable at follow up Week 24/Week 80 | 0.0 [0.00 to 13.23] | 6.1 [0.74 to 20.23]
  HBV-DNA <20000 IU/mL 1 year post-end of treatment: number analyzed (Participants) | 26 | 0
  HBV-DNA <20000 IU/mL 1 year post-end of treatment | 15.4 [4.36 to 34.87] |
  HBV-DNA <2000 IU/mL 1 year post-end of treatment: number analyzed (Participants) | 26 | 0
  HBV-DNA <2000 IU/mL 1 year post-end of treatment | 7.7 [0.95 to 25.13] |
  HBV-DNA Undetectable 1 year post-end of treatment: number analyzed (Participants) | 26 | 0
  HBV-DNA Undetectable 1 year post-end of treatment | 0.0 [0.00 to 13.23] |

7. Secondary Outcome: Change From Baseline in HBV DNA Levels in the Peg-INF-Alfa-2A (Treated) Arm
Description: This outcome measure presents HBV DNA levels measured at defined time points from baseline in the Peg-INF-Alfa-2A + Lamivudine or Entecavir arm.
Time Frame: Baseline, Week 8, 20, 32, 44, 56, Follow up Week 4 and 24
Population: The analysis population included participants from the Peg-INF-Alfa-2A arm, who received at least one dose of study medication of treated group. Only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir
Number analyzed (Participants) | 26
log10 IU/mL
  Baseline | 8.02 (0.93)
  Week 8: number analyzed (Participants) | 23
  Week 8 | 4.74 (1.01)
  Week 20: number analyzed (Participants) | 24
  Week 20 | 3.54 (0.81)
  Week 32: number analyzed (Participants) | 24
  Week 32 | 2.56 (0.84)
  Week 44: number analyzed (Participants) | 23
  Week 44 | 2.15 (0.70)
  Week 56: number analyzed (Participants) | 24
  Week 56 | 2.21 (0.90)
  Fu Week 4: number analyzed (Participants) | 20
  Fu Week 4 | 4.34 (2.65)
  Fu Week 24: number analyzed (Participants) | 21
  Fu Week 24 | 7.31 (1.99)

8. Secondary Outcome: Change From Baseline in HBV DNA Levels in the Untreated Control Participants
Description: This outcome measure presents HBV DNA levels measured at defined time points from baseline in the Untreated Control arm.
Time Frame: Baseline, Week 32, 56 and end of untreated observation (Week 80)
Population: The analysis population included participants from the Untreated Control arm. Only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Untreated Control Participants
Number analyzed (Participants) | 33
log10 IU/mL
  Baseline: number analyzed (Participants) | 32
  Baseline | 8.22 (1.07)
  Week 32: number analyzed (Participants) | 22
  Week 32 | 8.29 (0.97)
  Week 56: number analyzed (Participants) | 20
  Week 56 | 7.57 (1.96)
  Week 80: number analyzed (Participants) | 24
  Week 80 | 7.24 (2.58)

9. Secondary Outcome: Percentage of Participants With Combined Response for HBeAg Seroconversion (Defined as Loss of HBeAg and Presence of Anti-HBe) and HBV DNA Levels <20,000 IU/mL
Description: This endpoint measures the combined response for HBeAg Seroconversion and HBV DNA Levels <20,000 IU/mL at 24 weeks post-treatment (follow-up Week 24)/end of untreated observation (Week 80) and at 1 year post-end of treatment in the treated group. The HBeAg is defined as loss of HBeAg and presence of anti-HBe. The 95% Confidence Interval of response rate is calculated by Clopper-Pearson method.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants
Number analyzed (Participants) | 26 | 33
Percentage of Participants
  24 Weeks post-treatment/Week 80 | 0.0 [0.00 to 13.23] | 9.1 [1.92 to 24.33]
  1 year post-end of treatment: number analyzed (Participants) | 26 | 0
  1 year post-end of treatment | 7.7 [0.95 to 25.13] |

10. Secondary Outcome: Percentage of Participants With Combined Response for HBeAg Seroconversion (Defined as Loss of HBeAg and Presence of Anti-HBe) and HBV DNA Levels <2000 IU/mL
Description: This endpoint measures the combined response for HBeAg Seroconversion and HBV DNA Levels <2000 IU/mL at 24 weeks post-treatment (follow-up Week 24)/end of untreated observation (Week 80) and at 1 year post-end of treatment in the treated group. The HBeAg is defined as loss of HBeAg and presence of anti-HBe. The 95% Confidence Interval of response rate is calculated by Clopper-Pearson method.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants
Number analyzed (Participants) | 26 | 33
Percentage of Participants
  24 Weeks post-treatment/Week 80 | 0.0 [0.00 to 13.23] | 9.1 [1.92 to 24.33]
  1 year post-end of treatment: number analyzed (Participants) | 26 | 0
  1 year post-end of treatment | 7.7 [0.95 to 25.13] |

11. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to 24 weeks post-treatment/end of untreated observation (Week 80)
Population: The safety population included all participants who received at least one dose of study medication and had at least one post-baseline safety assessment. For untreated group, the safety population included all randomized participants who had at least one post-baseline safety assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants
Number analyzed (Participants) | 26 | 33
Percentage of Participants
  With at least one Non-Serious AE | 92.3 | 45.5
  With at least one Serious Adverse Event (SAE) | 0 | 3.0

12. Secondary Outcome: Percentage of Participants With AEs Leading to Dose Modification or Interruption
Description: This endpoint measures AEs and lab abnormalities leading to dose interruption or dose modification. Does modification included dose reduced, dose increased or drug interrupted. Adverse events included laboratory abnormalities reported as adverse events.
Time Frame: Baseline up to 24 weeks post-end of treatment
Population: The safety analysis population included all participants who received at least one dose of study medication and had at least one post-baseline safety assessment in the Peg-INF-Alfa-2A treated arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir
Number analyzed (Participants) | 26
Percentage of Participants | 23.0

13. Secondary Outcome: Serum Concentration of Peg-INF-Alfa-2A
Description: The serum concentration of Peg-INF-Alfa-2A was measured in picogram/milliliter.
Time Frame: At Weeks 12, 16, 20, 32, 44, 56
Population: The analysis population was the Peg-IFN-Alfa-2A + Lamivudine or Entecavir arm. The untreated arm did not receive any study medication. Only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir
Number analyzed (Participants) | 26
pg/mL
  Week 12 Predose: number analyzed (Participants) | 6
  Week 12 Predose | 8430 (6090)
  Week 16 Predose: number analyzed (Participants) | 8
  Week 16 Predose | 16300 (10100)
  Week 20 Predose: number analyzed (Participants) | 10
  Week 20 Predose | 13800 (8740)
  Week 32 Predose: number analyzed (Participants) | 11
  Week 32 Predose | 14900 (7710)
  Week 32 24-48h Post-dose: number analyzed (Participants) | 8
  Week 32 24-48h Post-dose | 22700 (6070)
  Week 32 72-96h Post-dose: number analyzed (Participants) | 8
  Week 32 72-96h Post-dose | 23000 (4900)
  Week 32 168h Post-dose: number analyzed (Participants) | 6
  Week 32 168h Post-dose | 19300 (5880)
  Week 44 Predose: number analyzed (Participants) | 9
  Week 44 Predose | 21900 (14200)
  Week 56 Predose: number analyzed (Participants) | 7
  Week 56 Predose | 25400 (13100)

ADVERSE EVENTS:
Time Frame: From Baseline up to 1 year post-end of treatment in the treated arm; From Baseline to end of untreated observation (Week 80) in the untreated group [up to clinical cut-off date 29 Jan 2020]
Description: The safety population included all participants who received at least one dose of study medication and had at least one post-baseline safety assessment. For untreated group, the safety population included all randomized participants who had at least one post-baseline safety assessment. Total # at Risk =0 in Other (Not Including Serious) Adverse Events section represents not reported data in consideration of participant re-identification.
Arm/Group | Peg-IFN-Alfa-2A + Lamivudine or Entecavir | Untreated Control Participants | Peg-INF-Alfa-2A Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/33 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/33 | 0/3
Other Adverse Events (participants affected / at risk) | 21/26 | 10/33 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peg-IFN-Alfa-2A + Lamivudine or Entecavir (N=26) | Untreated Control Participants (N=33) | Peg-INF-Alfa-2A Monotherapy (N=3)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peg-IFN-Alfa-2A + Lamivudine or Entecavir (N=26) | Untreated Control Participants (N=33) | Peg-INF-Alfa-2A Monotherapy (N=0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 2 (2) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 5 (11) | 0 (0) | 0 (0)
HYPERTHERMIA (General disorders) | 2 (3) | 0 (0) | 0 (0)
INJECTION SITE BRUISING (General disorders) | 2 (2) | 0 (0) | 0 (0)
PAIN (General disorders) | 3 (5) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 11 (21) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 2 (7) | 0 (0) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 14 (91) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 1 (1) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
In accordance with the recommendation from the DSMB, enrollment was stopped due to low efficacy and a changed benefit risk assessment. Enrolled participants were allowed to complete treatment and were followed up for 1 year after the end of treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT02263079/Prot_SAP_000.pdf